CLINICAL TRIAL: NCT05693935
Title: A Multinational, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study With an Open-Label, Long-Term Safety Phase to Evaluate the Efficacy, Safety, and Tolerability of Olanzapine for Extended-Release Injectable Suspension (TV-44749) for Subcutaneous Use as Treatment of Adult Patients With Schizophrenia
Brief Title: A Randomized, Double-Blind, Placebo-Controlled Study With an Open-Label, Long-Term Safety Phase to Evaluate the Efficacy and Safety of TV-44749 in Adults With Schizophrenia
Acronym: SOLARIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV44749-CNS-30096; 2022-001865-11 (EudraCT Number)
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Double-blind Period: Placebo (Placebo Comparator): Participants will receive placebo matched to TV-44749 subcutaneously (SC) once monthly over 8 weeks in double-blind period.
  Interventions: Drug: Placebo
- Double-blind Period: TV-44749 318 mg (Experimental): Participants will receive TV-44749 extended-release injectable suspension at a dose of 318 milligrams (mg) SC once monthly over 8 weeks in double-blind period.
  Interventions: Drug: TV-44749
- Double-blind Period: TV-44749 425 mg (Experimental): Participants will receive TV-44749 extended-release injectable suspension at a dose of 425 mg SC once monthly over 8 weeks in double-blind period.
  Interventions: Drug: TV-44749
- Double-blind Period: TV-44749 531 mg (Experimental): Participants will receive TV-44749 extended-release injectable suspension at a dose of 531 mg SC once monthly over 8 weeks in double-blind period.
  Interventions: Drug: TV-44749
- Open-label Period: Placebo to TV-44749 318 mg (Experimental): Participants who receive placebo during the double-blind period, will receive TV-44749 extended-release injectable suspension at a dose of 318 mg SC once monthly for up to 48 weeks in open-label period.
  Interventions: Drug: TV-44749
- Open-label Period: Placebo to TV-44749 425 mg (Experimental): Participants who receive placebo during the double-blind period, will receive TV-44749 extended-release injectable suspension at a dose of 425 mg SC once monthly for up to 48 weeks in open-label period.
  Interventions: Drug: TV-44749
- Open-label Period: Placebo to TV-44749 531 mg (Experimental): Participants who receive placebo during the double-blind period, will receive TV-44749 extended-release injectable suspension at a dose of 531 mg SC once monthly for up to 48 weeks in open-label period.
  Interventions: Drug: TV-44749

INTERVENTIONS:
Drug: TV-44749 — In Period 1, 2 monthly injections. In Period 2, up to 12 monthly injections
  Other Names: Olanzapine for Extended-Release Injectable Suspension
  Arms: Double-blind Period: TV-44749 318 mg; Double-blind Period: TV-44749 425 mg; Double-blind Period: TV-44749 531 mg; Open-label Period: Placebo to TV-44749 318 mg; Open-label Period: Placebo to TV-44749 425 mg; Open-label Period: Placebo to TV-44749 531 mg
Drug: Placebo — In Period 1, 2 monthly injections (Period 1 only)
  Arms: Double-blind Period: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of TV-44749 in adult participants with schizophrenia.

A key secondary objective is to further evaluate the efficacy of TV-44749 based on additional parameters in adult participants with schizophrenia.

A secondary objective is to evaluate the safety and tolerability of TV-44749 in adult participants with schizophrenia

Another secondary objective of this study is to evaluate the efficacy of TV-44749 from baseline to endpoint in Period 1 in adult participants with schizophrenia.

Total study duration is up to 61 weeks, and treatment duration is up to 56 weeks, with weekly visits during the first 8 weeks and then monthly in-clinic visits with weekly calls during the remainder of the treatment period.

DETAILED DESCRIPTION:
Participants with exacerbation of schizophrenia may be included. The study will be composed of 2 periods: Period 1 (the double-blind, placebo-controlled, efficacy and safety period) and Period 2 (open-label long term safety period). For each participant, the duration of Period 1 will be 8 weeks, and the duration of Period 2 will be up to 48 weeks. In Period 1, participants will be randomized to one of 3 TV-44749 treatment groups or a placebo group in a 1:1:1:1 ratio. All participants will be randomized again to one of the TV44749 treatment groups in a 1:1:1 ratio for Period 2. The end-of-treatment and follow-up visits will be at 4 and 8 weeks after the last dose of investigational medicinal product administration, respectively.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a current confirmed diagnosis of schizophrenia according to the DSM-5, for >1 year
* The participant has exacerbation of schizophrenia that started ≤8 weeks prior to screening and would benefit from psychiatric hospitalization or continued hospitalization for symptoms of schizophrenia.
* Participants who have received an antipsychotic treatment (other than clozapine) in the past year must have been responsive based on the investigator's judgment (and based on discussions with family members, caregivers, or healthcare professionals, as applicable).
* Body mass index between 18.0 and 40.0 kg/m2, inclusive, at the time of screening
* Women may be included only if they have a negative beta-human chorionic gonadotropin (β-HCG) test at screening and baseline
* Women of childbearing potential must agree not to try to become pregnant, and, unless they have exclusively same-sex partners, must agree to use a highly effective method of contraception prior to the first administration of IMP, and agree to continue the use of this method for the duration of the study, and for 70 days after the last dose of IMP
* The participant is in adequate health as determined by medical and psychiatric history, medical examination, electrocardiogram (ECG), serum chemistry, hematology, coagulation urinalysis, and serology.
* NOTE- Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* The participant has a current clinically significant DSM-5 diagnosis other than schizophrenia (has a primary current diagnosis other than schizophrenia or a comorbid diagnosis that is primarily responsible for the current symptoms and functional impairment).
* The participant has a known history of the following: (a) borderline personality disorder, antisocial personality disorder, or bipolar disorder; (b) traumatic brain injury causing ongoing cognitive difficulties, Alzheimer's disease, or another form of dementia, or any chronic organic disease of the central nervous system; and (c) intellectual disability of a severity that would impact ability to participate in the study.
* The participant was hospitalized for >14 days (with the exception of social or administrative hospitalization) in the current exacerbation episode prior to screening.
* The participant has a significant risk of violent behavior based on the participant's medical history or investigator's judgment.
* The participant has a significant risk of committing suicide based on the participant's medical history or C-SSRS, and the investigator's judgment.
* The participant is currently using an LAI antipsychotic or is still under the coverage period of the specific LAI at time of screening.
* The participant has taken clozapine or has received electroconvulsive therapy within the last 12 months prior to screening.
* The participant is currently receiving daily oral olanzapine at a dose >20 mg/day.
* The participant has current or a history of known hypersensitivity to olanzapine or any of the excipients of TV-44749 or the oral formulation of olanzapine.
* The participant has had a significant sedation or delirium after antipsychotic treatment according to medical and psychiatric history and as judged by the investigator or suffered from delirium due to a medical condition.
* The participant has a non-fasting glucose level of ≥200 mg/dL at screening
* The participant meets criteria for moderate to severe substance use disorder (based on DSM-5 criteria) within the past 6 months (excluding those related to caffeine or nicotine)
* NOTE- Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 675 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2025-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D LLC
Locations (82):
- United States (53):
  - Teva Investigational Site 15460, Bentonville, Arkansas
  - Teva Investigational Site 15465, Little Rock, Arkansas
  - Teva Investigational Site 15453, Rogers, Arkansas
  - Teva Investigational Site 15470, Anaheim, California
  - Teva Investigational Site 15459, Bellflower, California
  - Teva Investigational Site 15490, Garden Grove, California
  - Teva Investigational Site 15474, La Habra, California
  - Teva Investigational Site 15481, Lemon Grove, California
  - Teva Investigational Site 15491, Long Beach, California
  - Teva Investigational Site 15497, Los Angeles, California
  - Teva Investigational Site 15482, Los Angeles, California
  - Teva Investigational Site 15450, Orange, California
  - Teva Investigational Site 15455, Pico Rivera, California
  - Teva Investigational Site 15471, Riverside, California
  - Teva Investigational Site 15444, San Diego, California
  - Teva Investigational Site 15449, Santee, California
  - Teva Investigational Site 15461, Sherman Oaks, California
  - Teva Investigational Site 15483, Torrance, California
  - Teva Investigational Site 15457, Hialeah, Florida
  - Teva Investigational Site 15488, Hollywood, Florida
  - Teva Investigational Site 15498, Hollywood, Florida
  - Teva Investigational Site 15458, Hollywood, Florida
  - Teva Investigational Site 15489, Homestead, Florida
  - Teva Investigational Site 15452, Miami, Florida
  - Teva Investigational Site 15495, Miami, Florida
  - Teva Investigational Site 15446, Miami, Florida
  - Teva Investigational Site 15456, Miami, Florida
  - Teva Investigational Site 15479, Miami, Florida
  - Teva Investigational Site 15462, Miami, Florida
  - Teva Investigational Site 15496, Miami, Florida
  - Teva Investigational Site 15494, Miami Lakes, Florida
  - Teva Investigational Site 15467, Miami Lakes, Florida
  - Teva Investigational Site 15473, Miami Lakes, Florida
  - Teva Investigational Site 15484, Miami Springs, Florida
  - Teva Investigational Site 15477, West Palm Beach, Florida
  - Teva Investigational Site 15468, Atlanta, Georgia
  - Teva Investigational Site 15469, Decatur, Georgia
  - Teva Investigational Site 15500, Peachtree Corners, Georgia
  - Teva Investigational Site 15485, Chicago, Illinois
  - Teva Investigational Site 15480, Chicago, Illinois
  - Teva Investigational Site 15447, Shreveport, Louisiana
  - Teva Investigational Site 15442, Gaithersburg, Maryland
  - Teva Investigational Site 15466, Flowood, Mississippi
  - Teva Investigational Site 15487, St Louis, Missouri
  - Teva Investigational Site 15451, Marlton, New Jersey
  - Teva Investigational Site 15441, Charlotte, North Carolina
  - Teva Investigational Site 15454, Dayton, Ohio
  - Teva Investigational Site 15472, North Canton, Ohio
  - Teva Investigational Site 15478, Oklahoma City, Oklahoma
  - Teva Investigational Site 15448, Austin, Texas
  - Teva Investigational Site 15486, DeSoto, Texas
  - Teva Investigational Site 15464, Irving, Texas
  - Teva Investigational Site 15443, Richardson, Texas
- Bulgaria (12):
  - Teva Investigational Site 59210, Burgas
  - Teva Investigational Site 59203, Kazanlak
  - Teva Investigational Site 59208, Lovech
  - Teva Investigational Site 59214, Pleven
  - Teva Investigational Site 59207, Plovdiv
  - Teva Investigational Site 59215, Razgrad
  - Teva Investigational Site 59202, Rousse
  - Teva Investigational Site 59211, Sliven
  - Teva Investigational Site 59205, Sofia
  - Teva Investigational Site 59212, Sofia
  - Teva Investigational Site 59209, Veliko Tarnovo
  - Teva Investigational Site 59206, Vratsa
- China (10):
  - Teva Investigational Site 88052, Beijing
  - Teva Investigational Site 88044, Hangzhou
  - Teva Investigational Site 88060, Hefei
  - Teva Investigational Site 88055, Jining Shi
  - Teva Investigational Site 88068, Nanchang
  - Teva Investigational Site 88053, Shanghai
  - Teva Investigational Site 88054, Tianjin
  - Teva Investigational Site 88071, Wuhan
  - Teva Investigational Site 88072, Xinxiang
  - Teva Investigational Site 88064, Zhumadian
- Romania (4):
  - Teva Investigational Site 52124, Bucharest
  - Teva Investigational Site 52127, Bucharest
  - Teva Investigational Site 52123, Iași
  - Teva Investigational Site 52126, Iași
- Turkey (Türkiye) (3):
  - Teva Investigational Site 82058, Adapazarı
  - Teva Investigational Site 82059, Ankara
  - Teva Investigational Site 82057, Bursa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.

REFERENCES:
- [Derived] Cherniakov I, Wagner AM, Eshet R, Tiver R, Bibi D, Perlstein I, Kalmanczhelyi A, Sharon N, Cohen G, Ferderber K, Roberts J, Elgart A, Gutman D, Rabinovich-Guilatt L. Safety, Tolerability, and Pharmacokinetics of Subcutaneous Extended-Release Injectable Olanzapine in Patients with Schizophrenia and Schizoaffective Disorder. Clin Drug Investig. 2026 Feb 3. doi: 10.1007/s40261-025-01507-x. Online ahead of print. PMID 41632432
- [Derived] Perlstein I, Cherniakov I, Elgart A, Gomeni R, Gutman D, Merenlender Wagner A, Singh R. Population Pharmacokinetic Model-Based Dose Selection of Extended-Release Injectable Olanzapine (TV-44749) for Subcutaneous Use in Phase 3 Clinical Trial in Adults with Schizophrenia. J Clin Pharmacol. 2026 Jan;66(1):e70144. doi: 10.1002/jcph.70144. PMID 41496255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study comprised 2 periods: Period 1 (double-blind, placebo-controlled, efficacy and safety period [acute treatment phase]) and Period 2 (open-label safety period [long-term safety phase]).
Pre-assignment Details: Per planned analysis, the safety analysis was performed separately for Period 1 and for the integrated trial period. Integrated trial period included all participants who received 1 of the 3 TV-44749 treatments in Period 1 and all randomized participants to Period 2 who received at least 1 dose of TV-44749.
Groups:
- Placebo: Participants received placebo matched to TV-44749 subcutaneously (SC) once monthly over 8 weeks in double-blind period.
- TV-44749 318 mg: Participants received TV-44749 extended-release injectable suspension at a dose of 318 milligrams (mg) SC once monthly over 8 weeks in double-blind period and up to an additional 48 weeks in open-label period, for a total of 56 weeks.
- TV-44749 425 mg: Participants received TV-44749 extended-release injectable suspension at a dose of 425 mg SC once monthly over 8 weeks in double-blind period and up to an additional 48 weeks in open-label period, for a total of 56 weeks.
- TV-44749 531 mg: Participants received TV-44749 extended-release injectable suspension at a dose of 531 mg SC once monthly over 8 weeks in double-blind period and up to an additional 48 weeks in open-label period, for a total of 56 weeks.
- Placebo to TV-44749 318 mg: Participants who received placebo during the double-blind period, received TV-44749 extended-release injectable suspension at a dose of 318 mg SC once monthly for up to 48 weeks in open-label period.
- Placebo to TV-44749 425 mg: Participants who received placebo during the double-blind period, received TV-44749 extended-release injectable suspension at a dose of 425 mg SC once monthly for up to 48 weeks in open-label period.
- Placebo to TV-44749 531 mg: Participants who received placebo during the double-blind period, received TV-44749 extended-release injectable suspension at a dose of 531 mg SC once monthly for up to 48 weeks in open-label period.
Period: Double-blind Period (8 Weeks)
Arm/Group | Placebo | TV-44749 318 mg | TV-44749 425 mg | TV-44749 531 mg | Placebo to TV-44749 318 mg | Placebo to TV-44749 425 mg | Placebo to TV-44749 531 mg
Started (Full Analysis Set: all participants randomized to study arms in Period 1 regardless of the actual treatment the participants received.) | 168 | 169 | 169 | 169 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 167 | 164 | 168 | 168 | 0 | 0 | 0
Safety Analysis Set for Period 1 (All randomized participants who received at least 1 dose of TV-44749 or placebo. Participants were included in the treatment group corresponding to what they actually received.) | 167 | 163 (1 participant was randomized to receive TV-44749 318 mg but actually received TV-44749 531 mg.) | 168 | 169 (1 participant was randomized to receive TV-44749 318 mg but actually received TV-44749 531 mg.) | 0 | 0 | 0
Completed | 119 | 115 | 121 | 121 | 0 | 0 | 0
Not Completed | 49 | 54 | 48 | 48 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 4 | 2 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 26 | 35 | 31 | 33 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 4 | 6 | 4 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized But Not Treated | 1 | 5 | 1 | 1 | 0 | 0 | 0
Not completed — Other Than Specified | 11 | 5 | 8 | 7 | 0 | 0 | 0
Period: Open-label Period (48 Weeks)
Arm/Group | Placebo | TV-44749 318 mg | TV-44749 425 mg | TV-44749 531 mg | Placebo to TV-44749 318 mg | Placebo to TV-44749 425 mg | Placebo to TV-44749 531 mg
Started | 0 | 100 | 107 | 112 | 40 | 35 | 29
Received at Least 1 Dose of Study Drug | 0 | 100 | 106 | 112 | 40 | 35 | 29
Completed | 0 | 32 | 40 | 30 | 15 | 10 | 8
Not Completed | 0 | 68 | 67 | 82 | 25 | 25 | 21
Not completed — Adverse Event | 0 | 5 | 6 | 14 | 4 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 32 | 29 | 39 | 14 | 15 | 8
Not completed — Protocol Violation | 0 | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 17 | 19 | 17 | 3 | 5 | 4
Not completed — Lack of Efficacy | 0 | 1 | 2 | 1 | 0 | 1 | 2
Not completed — Randomized But Not Treated | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other Than Specified | 0 | 12 | 9 | 10 | 4 | 3 | 4

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all participants randomized to study arms in Period 1 regardless of the actual treatment the participants received.
Groups:
- Placebo: Participants received placebo matched to TV-44749 SC once monthly over 8 weeks in double-blind period.
- TV-44749 318 mg: Participants received TV-44749 extended-release injectable suspension at a dose of 318 mg SC once monthly over 8 weeks in double-blind period and up to an additional 48 weeks in open-label period, for a total of 56 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | TV-44749 318 mg | TV-44749 425 mg | TV-44749 531 mg | Total
Number analyzed (Participants) | 168 | 169 | 169 | 169 | 675
Age, Customized [Count of Participants; unit: Participants]
  18 - 30 years | 16 | 28 | 22 | 24 | 90
  >30 - 45 years | 86 | 59 | 65 | 64 | 274
  >45 - 65 years | 66 | 82 | 82 | 81 | 311
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 42 | 42 | 42 | 168
  Male | 126 | 127 | 127 | 127 | 507
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 38 | 34 | 32 | 132
  Not Hispanic or Latino | 139 | 130 | 135 | 135 | 539
  Unknown or Not Reported | 1 | 1 | 0 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 36 | 51 | 56 | 44 | 187
  Race: Black or African American | 121 | 116 | 106 | 119 | 462
  Race: Asian | 3 | 2 | 4 | 3 | 12
  Race: American Indian or Alaska Native | 2 | 0 | 1 | 1 | 4
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 2
  Race: Not reported | 0 | 0 | 0 | 2 | 2
  Race: Other | 5 | 0 | 1 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Double-blind Period: Change in the Positive and Negative Syndrome Scale (PANSS) Total Score From Baseline to Week 8
Description: The PANSS is a 30-item scale used to evaluate positive and negative symptoms of schizophrenia. The PANSS was used to identify the presence and severity of psychopathology symptoms, the relationship of these symptoms to one another, and the global psychopathology. Each item was scored on a 7-point scale ranging from 1 (absent) to 7 (extreme). The positive symptom scale includes 7 items with a maximum score of 49; the negative symptom scale includes 7 items with a maximum score of 49; and the general psychopathology scale includes 16 items with a maximum score of 112. The total score was the sum of 30-item scale, ranging from 30 (absent) to 210 (extreme), with a higher score indicating greater severity of symptoms. Least square (LS) mean was calculated using a repeated measures model with treatment, study visit, treatment visit interaction, stratification variables (sex and geographic region), age, and PANSS total score at baseline as covariates.
Time Frame: Baseline, Week 8
Population: Full Analysis Set included all participants randomized to study arms in Period 1 regardless of the actual treatment the participants received. 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Double-blind: Placebo: Participants received placebo matched to TV-44749 SC once monthly over 8 weeks in double-blind period.
- Double-blind: TV-44749 318 mg: Participants received TV-44749 extended-release injectable suspension at a dose of 318 mg SC once monthly over 8 weeks in double-blind period.
- Double-blind: TV-44749 425 mg: Participants received TV-44749 extended-release injectable suspension at a dose of 425 mg SC once monthly over 8 weeks in double-blind period.
- Double-blind: TV-44749 531 mg: Participants received TV-44749 extended-release injectable suspension at a dose of 531 mg SC once monthly over 8 weeks in double-blind period.
Arm/Group | Double-blind: Placebo | Double-blind: TV-44749 318 mg | Double-blind: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 165 | 163 | 166 | 165
units on a scale | -12.17 [-15.34 to -8.99] | -21.91 [-25.13 to -18.70] | -23.44 [-26.52 to -20.36] | -21.93 [-25.01 to -18.85]
Statistical Analysis 1: Comparison: Double-blind: Placebo vs Double-blind: TV-44749 318 mg; Mixed model for repeated measures fitted to 200 multiply imputed datasets generated in accordance with the estimand. Treatment group LS mean, 95% confidence intervals, and two-sided p values were pooled across imputations using Rubin's rules; Test type: Other; p < 0.0001, Mixed Models Analysis — p-value was adjusted for multiple comparisons (using Truncated Hochberg); LS Mean Difference = -9.75, 95% CI 2-sided [-13.60 to -5.89]
Statistical Analysis 2: Comparison: Double-blind: Placebo vs Double-blind: TV-44749 425 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Mixed Models Analysis — p-value was adjusted for multiple comparisons (using Truncated Hochberg); LS Mean Difference = -11.27, 95% CI 2-sided [-15.01 to -7.53]
Statistical Analysis 3: Comparison: Double-blind: Placebo vs Double-blind: TV-44749 531 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Mixed Models Analysis — p-value was adjusted for multiple comparisons (using Truncated Hochberg); LS Mean Difference = -9.76, 95% CI 2-sided [-13.50 to -6.02]

2. Secondary Outcome: Double-blind Period: Change in Clinical Global Impression-Severity (CGI-S) Scale Score From Baseline to Week 8
Description: The CGI-S is a 7-point scale that assess the participant's current severity of illness on a scale of 1 to 7, where 1=normal/not at all ill, 2=borderline mentally ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, and 7=among the most extremely ill patients. LS mean was calculated using a repeated measures model with treatment, study visit, treatment visit interaction, stratification variables (sex and geographic region), age, and CGI-S score at baseline as covariates.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Double-blind: Placebo | Double-blind: TV-44749 318 mg | Double-blind: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 165 | 163 | 166 | 165
units on a scale | -0.72 [-0.90 to -0.54] | -1.25 [-1.43 to -1.07] | -1.33 [-1.51 to -1.15] | -1.19 [-1.36 to -1.01]
Statistical Analysis 1: Comparison: Double-blind: Placebo vs Double-blind: TV-44749 318 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Mixed Models Analysis — p-value was adjusted for multiple comparisons (using Truncated Hochberg); LS Mean Difference = -0.53, 95% CI 2-sided [-0.75 to -0.31]
Statistical Analysis 2: Comparison: Double-blind: Placebo vs Double-blind: TV-44749 425 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Mixed Models Analysis — p-value was adjusted for multiple comparisons (using Truncated Hochberg); LS Mean Difference = -0.61, 95% CI 2-sided [-0.82 to -0.39]
Statistical Analysis 3: Comparison: Double-blind: Placebo vs Double-blind: TV-44749 531 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Mixed Models Analysis — p-value was adjusted for multiple comparisons (using Truncated Hochberg); LS Mean Difference = -0.47, 95% CI 2-sided [-0.68 to -0.25]

3. Secondary Outcome: Double-blind Period: Change in Personal and Social Performance Scale (PSP) Score From Baseline to Week 8
Description: The PSP is a clinician-rated instrument that measures personal and social functioning in participants with schizophrenia. The PSP is a 100-point single-item rating scale, divided into 10 equal intervals, where 0 (grossly impaired functioning) to 100 (excellent functioning). The score was based on the assessment of participant's functioning in 4 categories: 1) socially useful activities, including work and study; 2) personal and social relationships; 3) self-care; and 4) disturbing and aggressive behaviors. Higher scores represented better personal and social functioning, with ratings from 91 to 100 indicating more than adequate functioning, while scores under 30 indicating poor functioning that required intensive supervision. LS mean was calculated using a repeated measures model with treatment, study visit, treatment visit interaction, stratification variables (sex and geographic region), age, and PSP score at baseline as covariates.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Double-blind: Placebo | Double-blind: TV-44749 318 mg | Double-blind: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 165 | 163 | 166 | 165
units on a scale | 5.59 [3.14 to 8.04] | 10.31 [7.91 to 12.72] | 8.83 [6.44 to 11.22] | 10.59 [8.17 to 13.02]
Statistical Analysis 1: Comparison: Double-blind: Placebo vs Double-blind: TV-44749 318 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0011, Mixed Models Analysis — p-value was adjusted for multiple comparisons (using Truncated Hochberg); LS Mean Difference = 4.72, 95% CI 2-sided [2.05 to 7.40]
Statistical Analysis 2: Comparison: Double-blind: Placebo vs Double-blind: TV-44749 425 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0167, Mixed Models Analysis — p-value was adjusted for multiple comparisons (using Truncated Hochberg); LS Mean Difference = 3.24, 95% CI 2-sided [0.59 to 5.89]
Statistical Analysis 3: Comparison: Double-blind: Placebo vs Double-blind: TV-44749 531 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0007, Mixed Models Analysis — p-value was adjusted for multiple comparisons (using Truncated Hochberg); LS Mean Difference = 5.01, 95% CI 2-sided [2.35 to 7.66]

4. Secondary Outcome: Double-blind Period: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received the study drug without regard to possibility of causal relationship. The SAEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A TEAE was defined as an AE that occurred after the first dose of study drug was administered through end of the trial. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in the Reported AE section.
Time Frame: Baseline up to Week 8
Population: Safety Analysis Set for Period 1 included all randomized participants who received at least 1 dose of TV-44749 or placebo. Participants were included in the treatment group corresponding to what they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind: Placebo | Double-blind: TV-44749 318 mg | Double-blind: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 167 | 163 | 168 | 169
Participants
  Any TEAE | 84 | 112 | 117 | 126
  SAE | 3 | 4 | 1 | 2

5. Secondary Outcome: Integrated Study Period: Number of Participants With TEAEs and SAEs
Description: An AE was defined as any untoward medical occurrence in a participant who received the study drug without regard to possibility of causal relationship. The SAEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A TEAE was defined as an AE that occurred after the first dose of study drug was administered through end of the trial. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in the Reported AE section.
Time Frame: Baseline up to Week 60
Population: Safety Analysis Set for integrated study period included all participants in the safety analysis set of period 1 that received 1 of the 3 TV-44749 treatments groups and all randomized participants to Period 2 who received at least 1 dose of TV-44749. Participants were included in their randomized treatment groups regardless of the actual treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- Integrated Study Period: TV-44749 318 mg: Participants received TV-44749 extended-release injectable suspension at a dose of 318 mg SC once monthly over 8 weeks in double-blind period and up to an additional 48 weeks in open-label period, for a total of 56 weeks.
- Integrated Study Period: TV-44749 425 mg: Participants received TV-44749 extended-release injectable suspension at a dose of 425 mg SC once monthly over 8 weeks in double-blind period and up to an additional 48 weeks in open-label period, for a total of 56 weeks.
- Integrated Study Period: TV-44749 531 mg: Participants received TV-44749 extended-release injectable suspension at a dose of 531 mg SC once monthly over 8 weeks in double-blind period and up to an additional 48 weeks in open-label period, for a total of 56 weeks.
Arm/Group | Integrated Study Period: TV-44749 318 mg | Integrated Study Period: TV-44749 425 mg | Integrated Study Period: TV-44749 531 mg
Number analyzed (Participants) | 204 | 203 | 197
Participants
  Any TEAEs | 149 | 147 | 153
  SAEs | 15 | 8 | 13

6. Secondary Outcome: Double-blind Period: Change in PANSS Total Score From Baseline to Weeks 1, 2, and 4
Description: as for outcome 1
Time Frame: Baseline, Weeks 1, 2, and 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Double-blind: Placebo | Double-blind: TV-44749 318 mg | Double-blind: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 165 | 163 | 166 | 165
units on a scale
  Change at Week 1 | -5.74 [-8.09 to -3.39] | -7.54 [-9.86 to -5.21] | -7.29 [-9.61 to -4.96] | -6.22 [-8.53 to -3.91]
  Change at Week 2 | -7.95 [-10.50 to -5.40] | -11.02 [-13.54 to -8.50] | -11.25 [-13.75 to -8.75] | -10.05 [-12.54 to -7.55]
  Change at Week 4 | -9.40 [-12.16 to -6.65] | -15.27 [-18.03 to -12.51] | -15.91 [-18.61 to -13.21] | -14.74 [-17.43 to -12.05]

7. Secondary Outcome: Double-blind Period: Clinical Global Impression-Improvement (CGI-I) Scale Score at Weeks 4 and 8
Description: The CGI-I is a 7-point scale that permits a global evaluation of the participant's overall improvement in symptoms on a scale of 1 to 7, where 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse. LS mean was calculated using a repeated measures model with treatment, study visit, treatment visit interaction, stratification variables (sex and geographic region), age, and CGI-I score at baseline as covariates.
Time Frame: Weeks 4 and 8
Population: Full Analysis Set included all participants randomized to study arms in Period 1 regardless of the actual treatment the participants received. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind: Placebo | Double-blind: TV-44749 318 mg | Double-blind: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 146 | 131 | 152 | 150
units on a scale
  Week 4 | 3.42 (0.09) | 2.97 (0.09) | 3.00 (0.08) | 2.97 (0.08)
  Week 8: number analyzed (Participants) | 115 | 112 | 121 | 119
  Week 8 | 3.31 (0.10) | 2.64 (0.10) | 2.51 (0.10) | 2.56 (0.10)

8. Secondary Outcome: Double-blind Period: Change in CGI-S Scale Score From Baseline to Weeks 1, 2, and 4
Description: as for outcome 2
Time Frame: Baseline, Weeks 1, 2, and 4
Population: Full Analysis Set included all participants randomized to Period 1 regardless of the actual treatment the participants received. 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Double-blind: Placebo | Double-blind: TV-44749 318 mg | Double-blind: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 165 | 163 | 166 | 165
units on a scale
  Change at Week 1 | -0.27 [-0.41 to -0.13] | -0.33 [-0.47 to -0.19] | -0.33 [-0.47 to -0.19] | -0.23 [-0.37 to -0.10]
  Change at Week 2 | -0.42 [-0.57 to -0.27] | -0.56 [-0.72 to -0.41] | -0.59 [-0.74 to -0.44] | -0.48 [-0.63 to -.033]
  Change at Week 4 | -0.54 [-0.70 to -0.37] | -0.86 [-1.02 to -0.69] | -0.79 [-0.95 to -0.63] | -0.76 [-0.92 to -0.60]

9. Secondary Outcome: Double-blind Period: Patient Global Impression-Improvement (PGI-I) Scale Score at Weeks 2, 4, and 8
Description: The PGI-I scale is a 1-item participant-rated instrument that measures improvement of the participant's disease. The participant rated the perceived change in his/her condition in response to therapy on a scale of 1 to 7, where 1=very much better, 2=much better, 3=a little better, 4=no change, 5=a little worse, 6=much worse, 7=very much worse. LS mean was calculated using a repeated measures model with treatment, study visit, treatment visit interaction, stratification variables (sex and geographic region), age, and PGI-I score at baseline as covariates.
Time Frame: Weeks 2, 4, and 8
Population: Full Analysis Set included all participants randomized to Period 1 regardless of the actual treatment the participants received. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind: Placebo | Double-blind: TV-44749 318 mg | Double-blind: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 154 | 143 | 157 | 154
units on a scale
  Week 2 | 3.30 (0.11) | 2.95 (0.11) | 2.92 (0.11) | 3.16 (0.11)
  Week 4: number analyzed (Participants) | 143 | 131 | 149 | 147
  Week 4 | 3.24 (0.12) | 2.79 (0.12) | 2.92 (0.12) | 2.81 (0.12)
  Week 8: number analyzed (Participants) | 115 | 110 | 121 | 119
  Week 8 | 2.99 (0.13) | 2.46 (0.13) | 2.49 (0.12) | 2.43 (0.12)

10. Secondary Outcome: Double-blind Period: Change in Schizophrenia Quality of Life Scale (SQLS) Total Score From Baseline to Weeks 4 and 8
Description: The SQLS Revision 4 was administered to capture quality of life. The 33-item measure yields subscales pertaining to psychosocial (20 items) and cognition/vitality factors (13 items). Each item was scored on a 5-point scale (1 - never, 2 - rarely, 3 - sometimes, 4 - often, 5 - always). Individual domain and total scores were standardized by scoring algorithm from 0 (best health status) to 100 (worst health status) scale, with higher scores indicating comparatively lower quality of life.
Time Frame: Baseline, Weeks 4 and 8
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind: Placebo | Double-blind: TV-44749 318 mg | Double-blind: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 146 | 131 | 151 | 150
units on a scale
  Change at Week 4 | -5.63 (1.59) | -8.47 (1.62) | -7.16 (1.57) | -8.45 (1.58)
  Change at Week 8: number analyzed (Participants) | 115 | 110 | 121 | 119
  Change at Week 8 | -6.43 (1.79) | -10.42 (1.81) | -11.82 (1.75) | -12.08 (1.77)

11. Secondary Outcome: Double-blind Period: Change in PSP Score From Baseline to Week 4
Description: The PSP is a clinician-rated instrument that measures personal and social functioning in participants with schizophrenia. The PSP is a 100-point single-item rating scale, divided into 10 equal intervals, where 0 (grossly impaired functioning) to 100 (excellent functioning). The score was based on the assessment of participant's functioning in 4 categories: 1) socially useful activities, including work and study; 2) personal and social relationships; 3) self-care; and 4) disturbing and aggressive behaviors. Higher scores represented better personal and social functioning, with ratings from 91 to 100 indicating more than adequate functioning, while scores under 30 indicating functioning so poor that intensive supervision was required. LS mean was calculated using a repeated measures model with treatment, study visit, treatment visit interaction, stratification variables (sex and geographic region), age, and PSP score at baseline as covariates.
Time Frame: Baseline, Week 4
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Double-blind: Placebo | Double-blind: TV-44749 318 mg | Double-blind: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 165 | 163 | 166 | 165
units on a scale | 3.22 [1.02 to 5.42] | 6.14 [3.93 to 8.35] | 4.46 [2.30 to 6.62] | 4.88 [2.70 to 7.07]

12. Secondary Outcome: Double-blind Period: Number of Participants Receiving At Least 1 Concomitant Medication
Description: Concomitant medications included all medications taken while the participant was treated with the study drug. Any concomitant medication received by the participant for AEs was recorded on the case report form (CRF). Concomitant medications included: zolpidem, zopiclone, zaleplon, or diphenhydramine for insomnia; benztropine, trihexyphenidyl, or diphenhydramine for parkinsonian symptoms; propranolol and benzodiazepines for akathisia; lorazepam on an as-needed basis for indications other than akathisia (for example, anxiety); and antihistamine and anticholinergic drugs for agitation and insomnia.
Time Frame: Baseline up to Week 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind: Placebo | Double-blind: TV-44749 318 mg | Double-blind: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 167 | 163 | 168 | 169
Participants | 138 | 128 | 128 | 141

13. Secondary Outcome: Integrated Study Period: Number of Participants Receiving At Least 1 Concomitant Medication
Description: Concomitant medications included all medications taken while the participant was treated with the study drug. Any concomitant medication received by the participant for AEs was recorded on the CRF. Concomitant medications included: zolpidem, zopiclone, zaleplon, or diphenhydramine for insomnia; benztropine, trihexyphenidyl, or diphenhydramine for parkinsonian symptoms; propranolol and benzodiazepines for akathisia; lorazepam on an as-needed basis for indications other than akathisia (for example, anxiety); and antihistamine and anticholinergic drugs for agitation and insomnia.
Time Frame: Baseline up to Week 60
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Study Period: TV-44749 318 mg | Integrated Study Period: TV-44749 425 mg | Integrated Study Period: TV-44749 531 mg
Number analyzed (Participants) | 204 | 203 | 197
Participants | 148 | 142 | 156

14. Secondary Outcome: Double-blind Period: Change From Baseline to Week 8 in Abnormal Involuntary Movement Scale (AIMS) Total Score
Description: The AIMS is a 14-item scale that includes assessments of orofacial movements, extremity and truncal dyskinesia, examiner's judgment of global severity, subjective measures of awareness of movements and distress, and a yes/no assessment of problems concerning teeth and/or dentures. AIMS total score was calculated as a sum of items 1 through 7. Items 1 through 7 included facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). Each item was rated from 0 (none) to 4 (severe) The AIMS total score for Items 1-7 ranged from 0 (no dyskinesia) to 28 (severe dyskinesia) with a higher score indicating greater severity of the condition.
Time Frame: Baseline, Week 8
Population: Safety Analysis Set for Period 1 included all randomized participants who received at least 1 dose of TV-44749 or placebo. Participants were included in the treatment group corresponding to what they actually received. 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind: Placebo | Double-blind: TV-44749 318 mg | Double-blind: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 117 | 111 | 121 | 120
units on a scale | -0.1 (0.83) | -0.1 (0.81) | 0.0 (0.64) | 0.0 (0.50)

15. Secondary Outcome: Integrated Study Period: Change From Baseline to the End of Treatment (EOT) in AIMS Total Score
Description: as for outcome 14
Time Frame: Baseline, EOT (up to Week 56)
Population: Safety Analysis Set for integrated study period included all participants in the safety analysis set of period 1 that received 1 of the 3 TV-44749 treatments groups and all randomized participants to Period 2 who received at least 1 dose of TV-44749. Participants were included in their randomized treatment groups regardless of the actual treatment received. 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Integrated Study Period: TV-44749 318 mg | Integrated Study Period: TV-44749 425 mg | Integrated Study Period: TV-44749 531 mg
Number analyzed (Participants) | 107 | 99 | 100
units on a scale | -0.10 (1.213) | -0.10 (0.416) | -0.09 (0.793)

16. Secondary Outcome: Double-blind Period: Change From Baseline to Week 8 in Simpson-Angus Scale (SAS) Mean Score
Description: The SAS is a 10-item instrument for the assessment of neuroleptic-induced parkinsonism. The items on the scale include measurements of hypokinesia, rigidity, glabellar reflex, tremor, and salivation. Each item was rated on a 5-point scale (0 [normal] to 4 [severe]). The mean score was calculated by adding the individual item scores and dividing by 10, ranging from 0 (normal) to 4 (severe) with a higher score indicating greater severity of symptoms.
Time Frame: Baseline, Week 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind: Placebo | Double-blind: TV-44749 318 mg | Double-blind: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 116 | 111 | 121 | 119
units on a scale | -0.02 (0.142) | -0.02 (0.107) | 0.00 (0.065) | -0.01 (0.073)

17. Secondary Outcome: Integrated Study Period: Change From Baseline to the EOT in SAS Mean Score
Description: as for outcome 16
Time Frame: Baseline, EOT (up to Week 56)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Double-blind: TV-44749 531 mg: Participants received TV-44749 extended-release injectable suspension at a dose of 531 mg SC once monthly over 8 weeks in double-blind period and up to an additional 48 weeks in open-label period, for a total of 56 weeks.
Arm/Group | Integrated Study Period: TV-44749 318 mg | Integrated Study Period: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 107 | 99 | 100
units on a scale | -0.03 (0.154) | -0.01 (0.049) | -0.01 (0.077)

18. Secondary Outcome: Double-blind Period: Change From Baseline to Week 8 in Barnes Akathisia Rating Scale (BARS) Total Score
Description: The BARS is an instrument that assesses the severity of drug-induced akathisia. The BARS included 3 items for rating objective restless movements, subjective restlessness, and any subjective distress associated with akathisia that were scored on a 4-point scale of 0 (normal) to 3 (most severe) and summed up yielding a total score ranging from 0 (normal) to 9 (most severe). Higher scores indicated greater severity of akathisia.
Time Frame: Baseline, Week 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind: Placebo | Double-blind: TV-44749 318 mg | Double-blind: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 117 | 111 | 121 | 120
units on a scale | -0.1 (0.56) | -0.1 (0.66) | 0.0 (0.48) | -0.1 (0.50)

19. Secondary Outcome: Integrated Study Period: Change From Baseline to the EOT in BARS Total Score
Description: as for outcome 18
Time Frame: Baseline, EOT (up to Week 56)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Integrated Study Period: TV-44749 318 mg | Integrated Study Period: TV-44749 425 mg | Integrated Study Period: TV-44749 531 mg
Number analyzed (Participants) | 107 | 99 | 100
units on a scale | -0.1 (0.72) | -0.1 (0.52) | -0.1 (0.82)

20. Secondary Outcome: Double-blind Period: Number of Participants With Any Suicidal Ideation or Suicidal Behavior According to the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a questionnaire to assess suicidal ideation and suicidal behavior. Suicidal behavior was defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation was defined as a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent, any self-injurious behavior with no suicidal intent.
Time Frame: Baseline up to Week 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind: Placebo | Double-blind: TV-44749 318 mg | Double-blind: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 167 | 163 | 168 | 169
Participants
  No | 154 | 149 | 156 | 165
  Yes | 9 | 8 | 9 | 4
  Missing | 4 | 6 | 3 | 0

21. Secondary Outcome: Integrated Study Period: Number of Participants With Any Suicidal Ideation or Suicidal Behavior According to the C-SSRS
Description: as for outcome 20
Time Frame: Baseline up to Week 60
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Study Period: TV-44749 318 mg | Integrated Study Period: TV-44749 425 mg | Integrated Study Period: TV-44749 531 mg
Number analyzed (Participants) | 204 | 203 | 197
Participants
  No | 184 | 183 | 186
  Yes | 14 | 16 | 11
  Missing | 6 | 4 | 0

22. Secondary Outcome: Double-blind Period: Change From Baseline to Week 8 in Calgary Depression Scale for Schizophrenia (CDSS) Score
Description: The CDSS is specifically designed to assess the level of depression separate from the positive, negative, and extrapyramidal symptoms in schizophrenia. This clinician-administered instrument consisted of 9 items, each rated on a 4-point scale from 0 (absent) to 3 (severe) that are added together to form the CDSS depression total score for the participant ranging from 0 (absent) to 27 (severe) with higher scores indicating a higher severity of depression.
Time Frame: Baseline, Week 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind: Placebo | Double-blind: TV-44749 318 mg | Double-blind: TV-44749 425 mg | Double-blind: TV-44749 531 mg
Number analyzed (Participants) | 118 | 116 | 122 | 123
units on a scale | -1.1 (3.16) | -2.1 (3.95) | -1.7 (3.17) | -2.0 (3.77)

23. Secondary Outcome: Integrated Study Period: Change From Baseline to the EOT in CDSS Score
Description: as for outcome 22
Time Frame: Baseline, EOT (up to Week 56)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Integrated Study Period: TV-44749 318 mg | Integrated Study Period: TV-44749 425 mg | Integrated Study Period: TV-44749 531 mg
Number analyzed (Participants) | 107 | 99 | 101
units on a scale | -2.2 (4.08) | -1.6 (3.29) | -1.5 (3.72)

ADVERSE EVENTS:
Time Frame: Double-blind period: Baseline up to Week 8; Integrated study period: Baseline up to Week 60
Description: All-cause mortality data were collected and reported for all enrolled participants; and Serious and Non-serious adverse events data were collected and reported for all randomized participants who received at least 1 dose of TV-44749 or placebo.
Groups:
- Double Blind Period: Placebo: Participants received placebo matched to TV-44749 SC once monthly over 8 weeks in double-blind period.
- Double Blind Period: TV-44749 318 mg: Participants received TV-44749 extended-release injectable suspension at a dose of 318 mg SC once monthly over 8 weeks in double-blind period.
- Double Blind Period: TV-44749 425 mg: Participants received TV-44749 extended-release injectable suspension at a dose of 425 mg SC once monthly over 8 weeks in double-blind period.
- Double Blind Period: TV-44749 531 mg: Participants received TV-44749 extended-release injectable suspension at a dose of 531 mg SC once monthly over 8 weeks in double-blind period.
Arm/Group | Double Blind Period: Placebo | Double Blind Period: TV-44749 318 mg | Double Blind Period: TV-44749 425 mg | Double Blind Period: TV-44749 531 mg | Integrated Study Period: TV-44749 318 mg | Integrated Study Period: TV-44749 425 mg | Integrated Study Period: TV-44749 531 mg
All-Cause Mortality (participants affected / at risk) | 0/168 | 0/169 | 0/169 | 0/169 | 2/209 | 0/204 | 1/198
Serious Adverse Events (participants affected / at risk) | 3/167 | 4/163 | 1/168 | 2/169 | 15/204 | 8/203 | 13/197
Other Adverse Events (participants affected / at risk) | 38/167 | 82/163 | 99/168 | 98/169 | 105/204 | 113/203 | 113/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Blind Period: Placebo (N=167) | Double Blind Period: TV-44749 318 mg (N=163) | Double Blind Period: TV-44749 425 mg (N=168) | Double Blind Period: TV-44749 531 mg (N=169) | Integrated Study Period: TV-44749 318 mg (N=204) | Integrated Study Period: TV-44749 425 mg (N=203) | Integrated Study Period: TV-44749 531 mg (N=197)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug ineffective (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shoulder fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcoholic psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Psychotic symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 3 (3) | 8 (9)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Blind Period: Placebo (N=167) | Double Blind Period: TV-44749 318 mg (N=163) | Double Blind Period: TV-44749 425 mg (N=168) | Double Blind Period: TV-44749 531 mg (N=169) | Integrated Study Period: TV-44749 318 mg (N=204) | Integrated Study Period: TV-44749 425 mg (N=203) | Integrated Study Period: TV-44749 531 mg (N=197)
Constipation (Gastrointestinal disorders) | 6 (6) | 4 (4) | 8 (8) | 8 (10) | 7 (7) | 12 (12) | 9 (11)
Injection site erythema (General disorders) | 1 (1) | 12 (14) | 21 (25) | 15 (18) | 15 (19) | 24 (28) | 22 (27)
Injection site induration (General disorders) | 4 (6) | 18 (23) | 23 (29) | 23 (36) | 20 (30) | 27 (35) | 28 (43)
Injection site pain (General disorders) | 7 (7) | 14 (15) | 19 (25) | 17 (23) | 25 (26) | 25 (37) | 24 (34)
Injection site pruritus (General disorders) | 1 (1) | 9 (12) | 9 (9) | 11 (15) | 13 (35) | 12 (17) | 16 (26)
Injection site swelling (General disorders) | 1 (1) | 9 (12) | 10 (12) | 6 (7) | 11 (15) | 11 (14) | 8 (9)
Weight increased (Investigations) | 13 (13) | 49 (49) | 66 (66) | 58 (58) | 73 (74) | 78 (82) | 69 (74)
Headache (Nervous system disorders) | 11 (13) | 9 (9) | 14 (23) | 7 (9) | 9 (9) | 15 (25) | 8 (10)
Somnolence (Nervous system disorders) | 3 (3) | 16 (16) | 10 (11) | 13 (15) | 17 (18) | 11 (12) | 15 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT05693935/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT05693935/SAP_001.pdf